CLINICAL TRIAL: NCT02662374
Title: Efficacy of Two Different Oral Hygiene Regimens on the Incidence and Severity of Oral Mucositis in Patients Receiving Hematopoietic Stem Cell Transplantation - A Randomized Controlled Trial
Brief Title: Oral Hygiene Regimen in Patients on HCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Collaborators: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Sarah Ali Mubaraki, Post Graduate in Pediatric Dentistry, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RiyadhCDP
Record Dates: First submitted 2016-01-19; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Sodium Bicarbonate; Nystatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): 0.02% Chlorohexidine Gluconate: Mouth Rinse, 5ml, qid 3% Sodium Bicarbonate, Mouth Rinse, 5ml, qid Nystatin 10000U/ml : Mouth rinse, 5ml, qid
  Interventions: Drug: .02% Chlorohexidine Gluconate; Drug: 3% Sodium Bicarbonate; Drug: Nystatin 10000U/ml
- Group 1 (Experimental): 0.02% Chlorohexidine Gluconate: Mouth Rinse, 5ml, qid 3% Sodium Bicarbonate, Mouth Rinse, 5ml, qid Nystatin 10000U/ml : Mouth rinse, 5ml, qid Extra soft toothbrush, brushing with saline bd
  Interventions: Drug: .02% Chlorohexidine Gluconate; Drug: 3% Sodium Bicarbonate; Drug: Nystatin 10000U/ml; Device: Extra Soft Toothbrush
- Group 2 (Experimental): 0.02% Chlorohexidine Gluconate: Mouth Rinse, 5ml, qid 3% Sodium Bicarbonate, Mouth Rinse, 5ml, qid Nystatin 10000U/ml : Mouth rinse, 5ml, qid Supersaturated Calcium Phosphate Spray, 5ml qid
  Interventions: Drug: .02% Chlorohexidine Gluconate; Drug: 3% Sodium Bicarbonate; Drug: Nystatin 10000U/ml; Drug: Supersaturated Calcium Phosphate

INTERVENTIONS:
Drug: .02% Chlorohexidine Gluconate — 5ml of the drug in mouthwash form to be swished four times a day
  Other Names: Clorasept (ArRiyadh Pharmaceuticals, Riyadh, Saudi Arabia)
Drug: 3% Sodium Bicarbonate — 5ml of the drug in the form of a prepared solution to be swished four times a day
  Other Names: 3% Na2CO3
Drug: Nystatin 10000U/ml — 5ml of the drug in mouthwash form to be swished and swallowed four times a day
  Other Names: Mycostatin (Amman Pharmacuetical Corp. Amman, Jordan
Device: Extra Soft Toothbrush — To be moistened with 0.9% normal Saline and used twice daily to remove dental plaque
  Arms: Group 1
Drug: Supersaturated Calcium Phosphate — 5ml of the solution to be swished four times a day
  Other Names: Moistir (Kingswood laboratories Inc., Indianapolis IN USA)
  Arms: Group 2

SUMMARY:
Oral mucositis is one of the most common debilitating forms of mucositis that arise from high dose chemotherapy and radiotherapy. It is reported that almost 75% patients undergoing hematopoietic cell transplantation (HCT) develop oral mucositis at different levels of severity. The objective of this prospective study was to assess the efficacy of the addition of supersaturated calcium phosphate oral spray and the addition of an extra soft tooth brush to the basic OH in addition to the currently existing oral hygiene protocol regimen (0.2% Chlorhexidine Gluconate + 3% Sodium Bicarbonate+ Nystatin 100000 U/ml) in reducing the severity of oral mucositis among patients receiving chemotherapy for HCT.

60 patients receiving chemotherapy for HCT were randomly allocated to four groups of 15 patients each The oral mucositis was recorded according to WHO criteria and the progression of the oral mucositis was monitored from the day of admission (day

* 1) to the day of discharge (day 28). The absolute neutrophil count, platelet counts and salivary flow rate of all patients was recorded.

DETAILED DESCRIPTION:
This study will be prospective randomized case controlled study

Oral mucositis and oral hygiene protocol intervention:

45 patients admitted at King Faisal specialist hospital and Research Center in Riyadh for HCT and receiving chemotherapy regimen will be observed for the incidence and severity of oral mucositis.

Inclusion criteria:

* 3 to 16 years patients
* Male and female
* Allogeneic transplant
* Patient receiving conditioning regime

  * CYTOXAN, ATG, FLUDARABINE
  * BUSULPHAN/CYTOXAN/ATG WITH MTX
  * BUSULPHAN/CYTOXAN WITH MTX
  * FLUDARABINE/BUSULPHAN

Exclusion criteria:

* Patient age greater than 16 years and less than 3 years.
* Previous radiotherapy
* Had more than one graft.

Data Collection The child's age, gender, living area, type of disease, conditioning treatment protocol, absolute neutrophil count level, platelet count, use of opiate analgesics and patient reported outcome (pain, ability to eat, saliva flow rate and it is thickness) will be recorded.

Each patient will be examined once daily until discharge using the WHO criteria (see appendix I) At day -1

* All patient will receive an oral examination before chemo regimen or HCT started using the WHO oral health assessment form and the OM form as baseline for each patient.
* Start of the oral health protocol

Day 0, day 5, day10, day20, and day 25 Examination by tongue depressor and penlight to fill the OM form only and application of the oral hygiene protocol.

Oral health care protocol (OHCP):

Patients who fit the inclusion criteria will be randomly assigned to one of the following three groups Control group (15 patient) The control group will receive oral hygiene using the following protocol

* Chlorhexidine gluconate as a mouth wash 4 times daily
* Sodium bicarbonate mouth wash 4 times daily
* Patient can rinse by sterile water any time
* Nystatin will be administered 4 times.

Test group1 (15 patient)

* Twice a day oral prophylaxis by extra soft brush and water
* Chlorhexidine gluconate as a mouth wash 4 times daily
* Sodium bicarbonate mouth wash 4 times daily
* Patient can rinse by sterile water any time
* Nystatin will be administered 4 times.

Test group 2(15 patient)

* Supersaturated Calcium Spray 4 times daily
* Chlorhexidine gluconate as a mouth wash 4 times daily
* Sodium bicarbonate mouth wash 4 times daily
* Patient can rinse by sterile water any time
* Nystatin will be administered 4 times.

Test group 3(15 patient)

* Twice a day oral prophylaxis by extra soft brush and water Supersaturated Calcium Spray 4 times daily.
* Chlorhexidine gluconate as a mouth wash 4 times daily
* Sodium bicarbonate mouth wash 4 times daily
* Patient can rinse by sterile water any time
* Nystatin will be administered 4 times.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 16 years patients
* Male and female
* Allogeneic transplant
* Patient receiving conditioning regime

  * CYTOXAN, ATG, FLUDARABINE
  * BUSULPHAN/CYTOXAN/ATG WITH MTX
  * BUSULPHAN/CYTOXAN WITH MTX
  * FLUDARABINE/BUSULPHAN

Exclusion Criteria:

* Patient age greater than 16 years and less than 3 years.
* Previous radiotherapy
* Had more than one graft.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis Incidence | 28 days
  Presence of Oral Mucositis

SECONDARY OUTCOMES:
Oral Mucositis Severity | 28 Days
  Severity of Oral Mucositis measured using WHO criteria

CONTACTS AND LOCATIONS:
Overall Officials: abdullah R alshammery, PhD, Study Director — RiyadhCPD

IPD SHARING:
Plan to Share IPD: Undecided